CLINICAL TRIAL: NCT04814121
Title: Suxiao Jiuxin Pills in Microvascular Obstruction in Patients With Acute Coronary Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020KT1715
Record Dates: First submitted 2021-02-25; First posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Acute Coronary Syndrome
Keywords: Microvascular obstruction; Acute Coronary Syndrome; Percutaneous coronary intervention; Suxiao Jiuxin Pills
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suxiao Jiuxin Pills (Experimental): Suxiao Jiuxin Pills prescription (15 pills loading does, maintenance 6 pills each time, three times a day.) for 180 days
  Interventions: Drug: Suxiao Jiuxin Pills
- The placebo of Suxiao Jiuxin Pills (Placebo Comparator): The placebo of Suxiao Jiuxin Pills prescription (15 pills loading does, maintenance 6 pills each time, three times a day.) for 180 days
  Interventions: Drug: The placebo of Suxiao Jiuxin Pills

INTERVENTIONS:
Drug: Suxiao Jiuxin Pills — Suxiao Jiuxin Pills consists Rhizoma Ligustici (Chuan xiong) and Borneolum (Bing pian).
  Arms: Suxiao Jiuxin Pills
Drug: The placebo of Suxiao Jiuxin Pills — The placebo of Suxiao Jiuxin Pills is similar to Suxiao Jiuxin Pills in appearance, smell, and taste.
  Arms: The placebo of Suxiao Jiuxin Pills

SUMMARY:
Microvascular obstruction is the severe complication of percutaneous coronary intervention (PCI) in patients with acute coronary syndrome. Microvascular obstruction after PCI is often association with poor prognosis. Current treatments do not show improvement in prognosis of microvascular obstruction. Suxiao Jiuxin Pills (SXJX) was shown associated with a reduction in MACE, and an improvement of heart function and quality of life in acute coronary syndrome (ACS) patients with early PCI. To evaluate the effectiveness and safety of SXJX in microvascular obstruction after PCI, the investigators designed this study.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnosis of AMI, prepare for PCI reperfusion therapy;
* Between the ages of 18-75;
* Volunteer to participate in this study and have signed an informed consent form;
* Have a correct understanding of the significance of drug research, and have a good compliance with the observation and evaluation.

Exclusion Criteria:

* Not suitable for coronary intervention;
* With unstable hemodynamics;
* Platelet count<100×109;
* Suspected aortic dissection or acute pulmonary embolism;
* With mechanical complications;
* With uncontrolled acute left heart failure and pulmonary edema;
* With known bleeding history, active bleeding, bleeding constitution, or severe hemostatic and coagulation dysfunction;
* Meantain anticoagulants (such as warfarin or new anticoagulants);
* Severe liver and kidney insufficiency (Child-Pugh B and above, Cr>177μmol/L (2mg/dl) or eGFR<45ml/min/1.73m2);
* CTO, stent stenosis, or severe left main disease;
* History of coronary artery bypass graft surgery;
* Other pathophysiological conditions whose expected survival period is less than 1 year;
* Allergic history to Suxiao Jiuxin Pills;
* Pregnant or lactating women;
* Participating in other clinical studies;
* With other diseases that are not suitable for participating in clinical research.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline myocardial infarct size at 6 months | 3-5 days after PCI and 180±7 days
  MI size measure by CMR
Change from baseline incidence of microvascular obstruction at 6 months | 3-5 days after PCI and 180±7 days
  Incidence of Microvascular obstruction measure by CMR

SECONDARY OUTCOMES:
Change from baseline incidence of intramyocardial hemorrhagex at 6 months | 3-5 days after PCI and 180±7 days
  Incidence of intramyocardial hemorrhagex measure by CMR
Change from baseline incidence of area-at-risk at 6 months | 3-5 days after PCI and 180±7 days
  Incidence of area-at-risk measure by CMR
Change of ST segment in electrocardiogram | Baseline, immediately after PCI, 5-7 days after PCI, 30±7 days and 180±7 days
  Change of ST segment in electrocardiogram
Change of CK-MB | Baseline, immediately after PCI, 5-7 days after PCI, and 180±7 days
  CK-MB
Change of cTnI | Baseline, immediately after PCI, 5-7 days after PCI, and 180±7 days
  cTnI
Change of NT-proBNP | Baseline, immediately after PCI, 5-7 days after PCI, and 180±7 days
  NT-proBNP
Change of ejection fraction in echocardiography | Baseline, 3-5 days after PCI and 180±7 days
  Ejection fraction measure by echocardiography
Change of 6 Minute Walk Test | 3-5 days after PCI, 30±7 days and 180±7 days
  6MWT is used to assess aerobic capacity and endurance
Quantitative flow ratio | During the procedure
  Index measure by QFR
Incidence of MACCE | Through study completion, an average of 1 year
  Cardiac death, myocardial infarction, stent thrombosis, stroke or transient ischemic attack, urgent revascularization and re-hospitalization for heart failure
Incidence of complications of PCI | Up to 1 month
  Cardiac shock, heart failure, mechanical complications and arrhythmia
Incidence of bleeding event | Up to 6 months
  BARC Type 3 or 4
Incidence of stent restenosis | 180±7 days
  stent restenosis measure by CMR
Incidence of death event | Through study completion, an average of 1 year
  Any death
Change of Seattle Angina Questionnaire (SAQ) | baseline, 3-5 days after PCI, 30±7 days, 90±7 days and 180±7 days
  Seattle Angina Questionnaire (SAQ), the scale has 19 questions, value of each question is from 1 to 6, higher scores mean a better outcome.